CLINICAL TRIAL: NCT02884791
Title: Fibroblast Growth Factor 21 and Fructose Challenge in Humans
Brief Title: FGF21 and Fructose Challenge in Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Jody Dushay, Assistant Professor of Medicine, Beth Israel Deaconess Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2015P000381
Record Dates: First submitted 2016-03-23; First posted 2016-08-31 (Estimated); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Fasting
Keywords: FGF21; Fibroblast growth factor; fructose
MeSH Terms: conditions — Fasting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fasting (Healthy) (Experimental): Participation in this study involves fasting overnight, drinking a sweet beverage, and several blood draws through an IV line. Each subject may drink up to10 different sweet beverages, separated by 2 weeks.
  Interventions: Dietary Supplement: oral carbohydrate challenge
- Fasting (metabolic syndrome) (Experimental): Participation in this study involves fasting overnight, drinking a sweet beverage, and several blood draws through an IV line. Each subject may drink up to10 different sweet beverages, separated by 2 weeks.
  Interventions: Dietary Supplement: oral carbohydrate challenge

INTERVENTIONS:
Dietary Supplement: oral carbohydrate challenge — Participants will fast for 8 hours and then drink a beverage containing fructose.

SUMMARY:
The primary aim of this study is to examine the effect of acute ingestion of fructose on serum FGF21 levels. Subjects in this study will be lean volunteers and individuals with metabolic syndrome.

DETAILED DESCRIPTION:
Participation in this study involves fasting overnight, drinking a sweet beverage, and several blood draws through an IV line. Each subject may drink up to 10 different sweet beverages, separated by 2 weeks.

ELIGIBILITY:
Inclusion criteria for lean subjects:

* Men and women ages 18-60
* BMI 19-25 kg/m2; 19-23 for Asian subjects
* Stable weight (variation < 3 kg within 6 months of screening visit)
* Ability to give informed consent
* Ability to follow verbal and written instructions in English
* Use of medically approved form of contraception (monophasic oral contraception, intra uterine device, surgical sterilization or 2 combined barrier methods)

Specific exclusion criteria for lean subjects:

* Fasting blood glucose >100; 2 hr OGTT blood glucose >140
* Fasting triglycerides >150

Inclusion criteria for metabolic syndrome subjects:

3 or more of the following (based on joint scientific statement by Alberti et al, 2009:

* Fasting triglycerides >150 mg/dl (or on treatment for elevated triglycerides)
* HDL cholesterol <40 mg/dl in men or <50 mg/dl in women
* Blood pressure > 130/85 (or antihypertensive treatment in a subject with history of hypertension)
* Fasting BG >100
* Elevated waist circumference ** see below for race and ethnic specifications

Men Women

* Asian or Central, South or Native American > 90 cm > 80 cm
* Non-Asian, Non-Latino United States > 102 cm > 88 cm

General Exclusion criteria

* Type 1 or type 2 diabetes mellitus diagnosed according to American Diabetes Association criteria
* Coronary heart disease (history of myocardial infarction, unstable angina pectoris, or congestive heart failure)
* Uncontrolled hypertension (BP > 160/100 mmHg on or off antihypertensive medication)
* Marijuana or intravenous drug use
* Recent weight loss (> 3 kg within 6 months of the screening visit)
* Gastroparesis
* Inflammatory or irritable bowel disease
* Malignancy treated with chemotherapy within the past 3 years
* Depression or psychosis requiring hospitalization
* Renal insufficiency (creatinine clearance < 40 ml/min)
* Transaminases > 2x above the normal range
* Known liver disease
* Pregnancy within 6 months of the screening visit
* Lactation
* Failure to use medically approved contraceptive methods
* History of surgery for the treatment of obesity (gastric banding, gastric bypass, gastric stapling)
* Change in dose of thyroid hormone or antithyroidal medication within 3 months of screening visit
* History of alcohol abuse within the past 5 years
* Fructose intolerance

Exclusionary medications:

* Oral steroids
* Metformin
* Weight loss medications including nonprescription supplements

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-02 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
Change in Fibroblast Growth Factor 21 levels in human serum | 5 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No